CLINICAL TRIAL: NCT06677736
Title: Effect of Low-Level Laser Therapy on Salivary Toll Like Receptor- 4 Concentration of Periodontitis Patients: a Relation to Periodontal Inflammaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawda Saleh Saad Alashmawy (Other)
Responsible Party: Sponsor-Investigator, Rawda Saleh Saad Alashmawy, dentist, Misr University for Science and Technology
Organization: Misr University for Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022\0083
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Periodontal Disease
Keywords: inflamaging
MeSH Terms: conditions — Periodontal Diseases | interventions — Debridement; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- conventional scaling and debridement young age patient (Experimental): conventional scaling and debridement young age patient
  Interventions: Procedure: conventional scaling and debridement
- conventional scaling and debridement old age patient (Experimental): conventional scaling and debridement old age patient
  Interventions: Procedure: conventional scaling and debridement
- diode laser as adjunctive to scaling and debridement young age patient (Experimental): diode laser as adjunctive to scaling and debridement young age patient
  Interventions: Radiation: Diode laser as adjunctive to conventional scaling and debridement
- diode laser as adjunctive to scaling and debridement old age patient (Experimental): diode laser as adjunctive to scaling and debridement old age patient
  Interventions: Radiation: Diode laser as adjunctive to conventional scaling and debridement

INTERVENTIONS:
Procedure: conventional scaling and debridement — conventional scaling and debridement
  Arms: conventional scaling and debridement old age patient; conventional scaling and debridement young age patient
Radiation: Diode laser as adjunctive to conventional scaling and debridement — Diode laser as adjunctive to conventional scaling and debridement
  Arms: diode laser as adjunctive to scaling and debridement old age patient; diode laser as adjunctive to scaling and debridement young age patient

SUMMARY:
Effect of Low-Level Laser Therapy on Salivary Toll Like Receptor- 4 Concentration of Periodontitis Patients: A Relation to Periodontal Inflammaging

DETAILED DESCRIPTION:
Effect of Low-Level Laser Therapy on Salivary Toll Like Receptor- 4 Concentration of Periodontitis Patients: A Relation to Periodontal Inflammaging

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Aged below 40 or above 60.
3. Have at least 16 natural teeth excluding wisdom.
4. Provide informed consent and willingness to cooperate with study protocol.
5. Periodontitis stage II patients (23):

   * CAL from 3-4 mm.
   * Radiographic bone loss (15% to 33%).
   * No tooth loss due to periodontitis.
   * Maximum probing depth ≤ 5 mm, mostly horizontal bone loss

Exclusion Criteria:

* 1- Patients with any smoking habits 2- History of antibiotics in the previous three months. 3- Pregnant or lactating female. 4- Treatment with any systemic drug. 5- History of systemic disease. 6- Patients who received periodontal treatment in the last 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
Clinical attachment loss | Base line , follow up after 1 month , second follow up after 6 months
Gingival index | base line, follow up after 1 month, second follow up after 6 months
Toll like receptor - 4 | base line, follow up after 1 month, second follow up after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Misr university for science and technology, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided